CLINICAL TRIAL: NCT03594942
Title: Diagnostic Outcomes of Patients Presenting With Per Rectal Bleed in Surgical Departments of Services Hospital Lahore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Other Study IDs: s2
Record Dates: First submitted 2018-07-08; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Rectal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: procto sigmoidoscopy and biopsy if required — procto sigmoidoscopy of patients presenting with per rectal bleed will be carried out to locate the source of bleeding and biopsy if required.
  Other Names: colonoscopy, puch biopsy

SUMMARY:
It is a cross sectional study in which investigators will be recruiting patients of any sex above 12 years of age who will present to surgical outdoor with per rectal bleed. Investigators will then follow them through investigations to reach a certain diagnosis. Then investigators will be able to compile the data of diseases and their frequency, which are presenting with rectal bleed in their setup.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any sex above 12 years old
* patients with rectal bleed in OPD

Exclusion Criteria:

* Patient with acute rectal bleeding due to infection like dysentry
* Acute proctitis
* Acute colitis

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patintes will be from lahore city and adjacent areas
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of diseases in patients with rectal bleed | 6 weeks
  outcome of this study is to discover the frequency of diseases which are presenting with rectal bleed in our setup like hemorrhoids, anal fissure or rectal carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided